CLINICAL TRIAL: NCT05123729
Title: Community-Academic Partnerships to Address Disparities Within Rural and Urban Communities
Brief Title: Leveraging Social Innovation and Community-Engagement to Reduce Disparities in Outbreak Control Outcomes
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00099888; 40010565 (Other: National Institutes of Health)
Record Dates: First submitted 2021-11-15; First posted 2021-11-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Outbreak Investigation
MeSH Terms: interventions — Hospital Rapid Response Team

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crowdsourced campaign package: Disease prevention intervention developed using a crowdsourcing process.
  Interventions: Behavioral: Crowdsourced campaign package
- Rapid Response Team: Pilot a new hybrid training focused on contact tracing and case investigation.
  Interventions: Behavioral: Rapid Response Teams

INTERVENTIONS:
Behavioral: Crowdsourced campaign package — Disease prevention intervention developed using a crowdsourcing process.
  Groups: Crowdsourced campaign package
Behavioral: Rapid Response Teams — Pilot a new hybrid training focused on contact tracing and case investigation.
  Groups: Rapid Response Team

SUMMARY:
This study evaluates the impact of an intervention to increase viral transmission behaviors. The intervention will be developed through a crowdsourcing contest.

DETAILED DESCRIPTION:
NPIs that are community-driven and developed in collaboration with diverse partners, including community members, public health agencies, and researchers may offer an acceptable and effective approach to reducing viral transmission and addressing individual and socio-structural barriers that lead to worse virus-related outcomes. Our study goals are to use a crowdsourcing open call to identify exceptional ideas (e.g., messages, videos, communication and dissemination strategies) that promote disease testing and encourage the public to practice the 3 Ws, referred to as health-promotive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* specific zip codes in North Carolina (specific zip codes to be determined)
* no self-reported history of COVID-19 infection
* have not tested within the past 14 days

Exclusion Criteria:

* live outside of study area
* under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NC residents residing in urban and rural communities
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled as measured by enrollment log | Up to 3 years
  Number of participants enrolled as measured by enrollment log
Number of participants rating intervention as acceptable as measured by a post-intervention questionnaire | Up to 4 years
  Number of participants rating intervention as acceptable as measured by a post-intervention questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tiarney Ritchwood, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No